CLINICAL TRIAL: NCT00271778
Title: A Randomized Control Study of the Outcomes of Mastoidotympanoplasty Versus Tympanoplasty in Quiescent Tubotympanic Otitis Media
Brief Title: A Comparative Study of the Outcomes of 2 Surgical Procedures for Safe Type of Chronic Otitis Media
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karnataka Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M06b/2003-04
Record Dates: First submitted 2006-01-03; First posted 2006-01-04 (Estimated); Last update posted 2006-01-04 (Estimated); Status verified 2005-12

CONDITIONS: Chronic Otitis Media; Tubotympanic Disease
Keywords: Otitis media suppurative; surgery ear
MeSH Terms: conditions — Otitis Media, Suppurative | interventions — Tympanoplasty

INTERVENTIONS:
Procedure: mastoidotympanoplasty and tympanoplasty

SUMMARY:
Mastoidotympanoplasty is a recognised surgery that is performed for chronic otitis media. But whether mastoidectomy in addition to tympanoplasty is really necessary in each and every case of quiescent chronic otitis media still remains controversial. Hence this study has been undertaken to study the differences in the outcomes of the 2 surgical procedures performed for chronic otitis media in a randomized control design.

DETAILED DESCRIPTION:
Design: single blinded randomized control study. Setting: Tertiary referral medical college hospital. Sample size: 60. No of groups: 2 [30 cases in each group]. Group 1: Patients undergoing mastoidotympanoplasty. Group 2: Patients undergoing tympanoplasty only. No of strata: 3.

Outcomes:

1. Improvement of hearing
2. Closure of tympanic perforation
3. Recurrence of disease
4. external ear canal stenosis

Tools for measurement of outcomes [before and after surgery]:

1. Pure tone audiometry
2. Impedance audiometry
3. Otoendoscopy
4. External ear canal dimensions

ELIGIBILITY:
Inclusion Criteria:Chronic tubotympanic otitis media in quiescent phase with intact ossicular chain -

Exclusion Criteria:1. atticoantral otitis media 2. Specific otitis media 3. Sensorineural hearing loss 4. Fixed/Dislocated ossicular chain 5. Uncorrectable disease focus in nose/throat 6. Chronic otitis media in active phase 7. Chronic otitis media with complications 8. Extensive unresectable tympanosclerosis

-

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2003-07; Study Completion 2006-06

PRIMARY OUTCOMES:
Pure tone audiometry
Impedance audiometry
Otoendoscopy
External ear canal dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Vikram K Bhat, MS, DNB., Principal Investigator — Karnataka Institute of Medical Sciences, Hubli, India; Khaja Naseeruddin, MS, DLO., Study Director — Vijayanagar Institute of Medical Sciences, Bellary, India
Locations (1):
- Department of ENT, KIMS, Hubli, Karnataka, India